CLINICAL TRIAL: NCT05939986
Title: Virtual Reality Exposure Therapy for Fear of Flying: Protocol for a Randomized Controlled Trial
Brief Title: A Protocol for a Virtual Reality Exposure Therapy for Fear of Flying.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, José María Ribé Viñes, Principal Investigator, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2926863
Record Dates: First submitted 2023-05-25; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Aerophobia; Virtual Reality Exposure Therapy; Randomized Controlled Trial; Anxiety
Keywords: Virtual Reality; Fear of Flying; Exposure; Vibrotactile Cues; Anxiety; Presence
MeSH Terms: conditions — Aerophobia; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of three intervention arms, namely the VRET with multimodal feedback (visual, auditory, and vibrotactile; VRET-M), the VRET with bimodal feedback (visual and auditory; VRET-B), or the imagery exposure treatment (IET).
Masking Description: Not-blinded study protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multimodal Virtual Reality Exposure Treatment (VRET-M) (Experimental): VRET with multimodal feedback including visual, auditory and vibrotactile cues.
  Interventions: Behavioral: Virtual reality-based exposure treatment with bimodal feedback (VRET-B); Behavioral: Imagery exposure treatment (IET)
- Bimodal Virtual Reality Exposure Treatment (VRET-B) (Active Comparator): VRET with bimodal feedback including visual and auditory cues.
  Interventions: Behavioral: Virtual reality-based exposure treatment with multimodal feedback (VRET-M); Behavioral: Imagery exposure treatment (IET)
- Imagery Exposure Treatment (IET) (Active Comparator): Imagery exposure treatment without sensory cues.
  Interventions: Behavioral: Virtual reality-based exposure treatment with multimodal feedback (VRET-M); Behavioral: Virtual reality-based exposure treatment with bimodal feedback (VRET-B)

INTERVENTIONS:
Behavioral: Virtual reality-based exposure treatment with multimodal feedback (VRET-M) — The VRET-M group will experience visual, auditive and vibrotactile cues in the exposure sessions.
  Arms: Bimodal Virtual Reality Exposure Treatment (VRET-B); Imagery Exposure Treatment (IET)
Behavioral: Virtual reality-based exposure treatment with bimodal feedback (VRET-B) — The VRET-B group will experience visual and auditive cues in the exposure sessions.
  Arms: Imagery Exposure Treatment (IET); Multimodal Virtual Reality Exposure Treatment (VRET-M)
Behavioral: Imagery exposure treatment (IET) — The IET group will experience its own subjective imagined environment without any external stimulation.
  Arms: Bimodal Virtual Reality Exposure Treatment (VRET-B); Multimodal Virtual Reality Exposure Treatment (VRET-M)

SUMMARY:
This study aims to assess whether adding vibrotactile stimulation to visual and auditory stimulation increases the efficacy of VRET for FoF treatment. Eighty-four participants (18-65 years old) will be assigned to one of three intervention arms, namely the VRET with multimodal feedback (visual, auditory, and vibrotactile; VRET-M), the VRET with bimodal feedback (visual and auditory; VRET-B), or the imagery exposure treatment (IET) without sensory feedback. FoF-related symptoms (primary outcomes) will be measured administering the Fear of Flying Questionnaire-II (QPV-II), the Fear of Flying Scale (FFS), and the Visual Analogic Scale (VAS-A) before and after eight sessions of treatment, and at six- and 12-month follow-ups. Anxiety and the sense of presence experienced during exposure sessions (secondary outcome measures: VAS-A and VAS-P) will also be assessed. It is expected that participants in the VRET-M group will report a further reduction of FoF-related symptomatology after the treatment and at follow-ups compared to participants in the VRET-B and IET groups. Likewise, participants in the VRET-M group are expected to show higher sense of presence levels during exposure sessions in comparison to participants in the VRET-B and IET groups. It is expected that the IET group will report the lowest level of sense of presence and the poorest outcome after treatment and at follow-ups.

DETAILED DESCRIPTION:
Participants who meet the inclusion criteria will be invited to participate in the initial treatment session. They will be also required to purchase a flight ticket during the six months after the end of the treatment. Participants will be treated weekly for eight individual sessions. While the first two sessions involve preparation and training, exposure will be conducted between the third and eighth session. The exposure sessions' structure and content will be the same in all conditions. Nevertheless, the VRET-M group will experience vibrotactile cues, while the VRET-B group will not. Furthermore, the IET group will experience its own subjective imagined environment without any external stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet the Diagnostic and Statistical Manual of Mental Disorders (DSM-5, American Psychiatric Association, APA, 2013) criteria for FoF.

Exclusion Criteria:

* Individuals with a diagnosis of panic disorder, obsessive-compulsive disorder, or psychotic disorder who have received psychotherapy for their FoF, have been taking prescribed medication for their FoF, or have experienced cardiorespiratory disease or an epilepsy attack will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2023-10-15 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Fear of Flying (FoF). Administering the Fear of Flying Questionnaire-II (QPV-II) and the Fear of Flying Scale (FFS). | Before the exposure treatment.
  To what extend I feel fear about flying by plane? The QPV-II is rated from on a 10-point scale (0 = absence of anxiety, 10 = extreme anxiety) with scores ranging from 0 to 300. The FFS is rated on a 5-point scale (0 = not at all, 4 = very much), with scores ranging from 0 to 84.
Fear of Flying (FoF). Administering the Fear of Flying Questionnaire-II (QPV-II) and the Fear of Flying Scale (FFS). | After eight sessions of treatment during eight weeks.
  To what extend I feel fear about flying by plane? The QPV-II is rated from on a 10-point scale (0 = absence of anxiety, 10 = extreme anxiety) with scores ranging from 0 to 300. The FFS is rated on a 5-point scale (0 = not at all, 4 = very much), with scores ranging from 0 to 84.
Fear of Flying (FoF). Administering the Fear of Flying Questionnaire-II (QPV-II) and the Fear of Flying Scale (FFS). | At 6 months follow-up after treatment termination.
  To what extend I feel fear about flying by plane? The QPV-II is rated from on a 10-point scale (0 = absence of anxiety, 10 = extreme anxiety) with scores ranging from 0 to 300. The FFS is rated on a 5-point scale (0 = not at all, 4 = very much), with scores ranging from 0 to 84.
Fear of Flying (FoF). Administering the Fear of Flying Questionnaire-II (QPV-II) and the Fear of Flying Scale (FFS). | At 12 months follow-up after treatment termination.
  To what extend I feel fear about flying by plane? The QPV-II is rated from on a 10-point scale (0 = absence of anxiety, 10 = extreme anxiety) with scores ranging from 0 to 300. The FFS is rated on a 5-point scale (0 = not at all, 4 = very much), with scores ranging from 0 to 84.
Anxiety. Administering a Visual Analogue Scale (VAS-A). | Before the exposure treatment.
  To what extend I feel anxious about flying by plane? measured from 0 (absence of anxiety) to 10 (extreme anxiety).
Anxiety. Administering a Visual Analogue Scale (VAS-A). | After eight sessions of treatment during eight weeks.
  To what extend I feel anxious about flying by plane? measured from 0 (absence of anxiety) to 10 (extreme anxiety).
Anxiety. Administering a Visual Analogue Scale (VAS-A). | At 6 months follow-up after treatment termination.
  To what extend I feel anxious about flying by plane? measured from 0 (absence of anxiety) to 10 (extreme anxiety).
Anxiety. Administering a Visual Analogue Scale (VAS-A). | At 12 months follow-up after treatment termination.
  To what extend I feel anxious about flying by plane? measured from 0 (absence of anxiety) to 10 (extreme anxiety).

SECONDARY OUTCOMES:
Anxiety. Administering a Visual Analogue Scale (VAS-A). | Before each exposure session.
  To what extend I feel anxious now? measured from 0 (absence of anxiety) to 10 (extreme anxiety).
Anxiety. Administering a Visual Analogue Scale (VAS-A). | Every 2 minutes during each exposure session of 60 minutes.
  To what extend I feel anxious now? measured from 0 (absence of anxiety) to 10 (extreme anxiety).
Anxiety. Administering a Visual Analogue Scale (VAS-A). | After eight sessions of treatment during eight weeks.
  To what extend I feel anxious now? measured from 0 (absence of anxiety) to 10 (extreme anxiety).
Sense of Presence. Administering the Visual Analogue Scale (VAS-P). | Every 2 minutes during each exposure session of 60 minutes.
  To what extend I feel present now? measured from 0 (absence of sense of presence) to 10 (extreme sense of presence).

CONTACTS AND LOCATIONS:
Overall Officials: José MR Gutiérrez Maldonado, PhD, Study Director — Senior PhD Supervisor
Locations (1):
- Faculty of Psychology. Universitat de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Gerwen LJ, Spinhoven P, Van Dyck R. Behavioral and cognitive group treatment for fear of flying: a randomized controlled trial. J Behav Ther Exp Psychiatry. 2006 Dec;37(4):358-71. doi: 10.1016/j.jbtep.2006.05.002. Epub 2006 Jul 7. PMID 16828460
- [Result] Rothbaum BO, Hodges L, Anderson PL, Price L, Smith S. Twelve-month follow-up of virtual reality and standard exposure therapies for the fear of flying. J Consult Clin Psychol. 2002 Apr;70(2):428-32. doi: 10.1037//0022-006x.70.2.428. PMID 11952201